CLINICAL TRIAL: NCT05866159
Title: The Effect of Kinesio Tape on Back-Specific Body Perception, Pain, Functional Status, and Physical Activity Level in Patients With Chronic Low Back Pain
Brief Title: Effects of Kinesio Tape on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Hakan AKKAN, PhD, PT, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KutahyaHSU-003
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain
Keywords: functional disability; pain; kinesiotape; physical activity
MeSH Terms: conditions — Low Back Pain; Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: comparing the use of kinesiotape for the treatment of back-specific body image, pain, functional disability, and physical activity of individuals with non-specific CLBP to sham-taping
Who Masked: Participant, Outcomes Assessor
Masking Description: A double-blinded design will be conducted to assess the effectiveness of kinesio versus sham tape, as patients cannot distinguish between the two.
  The assessment of back-specific body perception, which is the primary outcome, will be conducted by an assessor unaware of the treatment allocation prior to treatment, as well as on days 3 and 7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Intervention (Experimental): The experimental group will receive double-sided I-shaped kinesiotape. The tape will be applied from the sacroiliac joint to the thoracic 12th vertebrae, with a 10-15% tension. During the application, the participant will be positioned in maximum torso flexion.
  Interventions: Other: Kinesiotape using Rocktape®
- Control Intervention (Sham Comparator): For the sham group, the kinesiotape will be applied horizontally to the center of the painful area in the lumbar region without any tension (at 0%).
  Interventions: Other: Sham taping

INTERVENTIONS:
Other: Kinesiotape using Rocktape® — Kinesiotape using Rocktape® on day one by a physiotherapist who has experienced more than five years. If possible, the taping will be left for seven days.
  Arms: Experimental Intervention
Other: Sham taping — sham taping with Rocktape®, with no tension.
  Arms: Control Intervention

SUMMARY:
This clinical trial aims to examine kinesiotape's (KT) short-term effect on individuals with nonspecific chronic LBP (CLBP), including back-specific body perception, pain, functional disability, and physical activity. The hypothesis is that applying KT to the lumbar spine would improve back-specific body perception, reduce pain and functional disability, and increase physical activity in individuals with CLBP compared to the sham-taping group.

DETAILED DESCRIPTION:
Low back pain (LBP) is prevalent and the leading cause of disability worldwide. In addition, it is often associated with psychological, social, and physical factors that can impact one's ability to function, participate in society, maintain job satisfaction, and socioeconomic status. Therefore, managing it requires a significant amount of healthcare resources. Maladaptive body image and maladaptive beliefs are among the conditions that can be targeted during treatment as they may contribute to the chronicity of LBP.

This clinical trial aims to examine kinesiotape's (KT) short-term effect on individuals with nonspecific chronic LBP (CLBP), including back-specific body perception, pain, functional disability, and physical activity. The hypothesis is that applying KT to the lumbar spine would improve back-specific body perception, reduce pain and functional disability, and increase physical activity in individuals with CLBP compared to the sham-taping group.

ELIGIBILITY:
Inclusion Criteria:

* ability to speak and write Turkish fluently
* have been experiencing low back pain for at least 3 months
* have a pain severity score of ≥4 on the visual analog scale

Exclusion Criteria:

* had significant spinal surgery in the past (fusion or discectomy), spinal surgery within the last six months,
* a diagnosis of a serious spinal condition (such as cancer, inflammatory arthropathy, or vertebral fracture),
* skin allergy to KT or pre-existing skin lesion or infection
* a neurological disease,
* is currently pregnant,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Change in The Fremantle Back Awareness Questionnaire (FreBAQ) on day 1 and day 7 (in points) | day 1 before the start of the kinesiotaping, day 3, and day 7
  The Fremantle Back Awareness Questionnaire (FreBAQ) is a tool used to measure a patient's perception of their back. It consists of nine questions rated on a five-point scale, ranging from "0=never" to "4=always".

SECONDARY OUTCOMES:
Change in Pain Intensity (VAS) on day 0 and day 7 (in millimeters) | day 1 before the start of the kinesiotaping, day 3, and day 7
  Patients will score their low-back pain intensity over the past week on a horizontal 10 cm line with descriptive anchors at each end, such as on the right, "no pain" to the left, and "extreme pain."
Change in The Roland-Morris Disability Questionnaire (RMDQ) on day 1 and day 7 (in points) | day 1 before the start of the kinesiotaping, day 3, and day 7
  The RMDQ evaluates self-reported physical disability resulting from low back pain. The RMDQ questionnaire consists of 24 items. Each item is scored as "0" if left blank or "1" if endorsed. The total RMQ score ranges from 0 to 24, with higher scores indicating more pain-related disability.
Change in The International Physical Activity Questionnaire - Short Form (IPAQ-SF) on day 1 and day 7 (in MET min/wk) | day 1 before the start of the kinesiotaping, day 3, and day 7
  The IPAQ was developed to assess physical activity internationally. There are two versions of the International Physical Activity Questionnaire (IPAQ): the long form with 31 items (IPAQ-LF) and the short form with nine items (IPAQ-SF). The IPAQ-SF measures activity in four different intensity levels, including 1)vigorous activities, 2) moderate activities, 3) walking, and 4) sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Akkan, PhD, PT, Principal Investigator — Kütahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Sanchez AM, Lara-Palomo IC, Mataran-Penarrocha GA, Fernandez-Sanchez M, Sanchez-Labraca N, Arroyo-Morales M. Kinesio Taping reduces disability and pain slightly in chronic non-specific low back pain: a randomised trial. J Physiother. 2012;58(2):89-95. doi: 10.1016/S1836-9553(12)70088-7. PMID 22613238
- [Background] Koroglu F, Colak TK, Polat MG. The effect of Kinesio(R) taping on pain, functionality, mobility and endurance in the treatment of chronic low back pain: A randomized controlled study. J Back Musculoskelet Rehabil. 2017 Sep 22;30(5):1087-1093. doi: 10.3233/BMR-169705. PMID 28968232
- [Background] Luz Junior MA, Sousa MV, Neves LA, Cezar AA, Costa LO. Kinesio Taping(R) is not better than placebo in reducing pain and disability in patients with chronic non-specific low back pain: a randomized controlled trial. Braz J Phys Ther. 2015 Nov-Dec;19(6):482-90. doi: 10.1590/bjpt-rbf.2014.0128. Epub 2015 Oct 9. PMID 26647750
- [Background] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235
- [Background] Erol E, Yildiz A, Yildiz R, Apaydin U, Gokmen D, Elbasan B. Reliability and Validity of the Turkish Version of the Fremantle Back Awareness Questionnaire. Spine (Phila Pa 1976). 2019 May 1;44(9):E549-E554. doi: 10.1097/BRS.0000000000002909. PMID 30325886
- [Background] Macedo LB, Richards J, Borges DT, Melo SA, Brasileiro JS. Kinesio Taping reduces pain and improves disability in low back pain patients: a randomised controlled trial. Physiotherapy. 2019 Mar;105(1):65-75. doi: 10.1016/j.physio.2018.07.005. Epub 2018 Jul 26. PMID 30348455